CLINICAL TRIAL: NCT02695043
Title: Multimedia Multicultural Educational Program for Traumatic Brain Injury
Brief Title: MMEPT for Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00356
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMPET Group (Experimental): This group of subjects will be comprised of a subset of culturally diverse patients admitted to the Bellevue the Traumatic Brain Injury Unit at Bellevue. Treatment will focus on improving awareness and comprehension of TBI and its long-term consequences, fostering increased trust in the TBI rehabilitation team, and conveying the importance of continued TBI follow up to maximize recovery.
  Interventions: Behavioral: Multimedia Multicultural Educational Program for TBI (MMEPT)
- Control Group (Active Comparator): The Control Group will be comprised of equally diverse subset of patients who will receive Standard of Care Treatment.
  Interventions: Behavioral: RRTBIMS

INTERVENTIONS:
Behavioral: RRTBIMS — TBI patients discharged from Bellevue inpatient rehabilitation and enrolled in the Rusk Rehabilitation Traumatic Brain Injury Model System (RRTBIMS)
  Arms: Control Group
Behavioral: Multimedia Multicultural Educational Program for TBI (MMEPT)
  Arms: MMPET Group

SUMMARY:
The primary purpose of this research is to increase adherence to outpatient rehabilitation of chronically underserved individuals with traumatic brain injury (TBI). The intervention will be a TBI rehabilitation-focused education tool suitable for use with a wide variety of patients, including those with poor literacy skills and those with Limited English Proficiency (LEP), hereafter referred to as the Multimedia Multicultural Educational Program for TBI (MMEPT).

ELIGIBILITY:
Inclusion Criteria:

* A medically documented (e.g., EMS report, hospital record, physician record) TBI as a result of a blow to the head requiring admission to an acute inpatient rehabilitation unit, meeting at least one of the following criteria for moderate to severe TBI:

  1. PTA > 24 hours
  2. Trauma related intracranial neuroimaging abnormalities
  3. Loss of consciousness exceeding 30 minutes
  4. GCS in emergency department of less than 13 (unless due to intubation, sedation or intoxication)
* Proficient in Chinese (Mandarin or Cantonese), Spanish or English,
* Willing to engage in the MMEPT and complete questionnaires,
* Agreeing to participate (i.e., completion of informed consent and HIPAA documents).

Exclusion Criteria:

* Preferred language (language with greatest proficiency) other than English, Chinese or Spanish,
* In minimally conscious or vegetative state,
* Significant symptoms of receptive aphasia, and
* Any acute medical condition that, in the investigator's opinion, makes the person unsuitable or unable to participate. Participants enrolled in the study who are ultimately not discharged to the community at the completion of acute inpatient rehabilitation will be removed from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Difference in Rate of Retention | Up to One Week

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bushnik, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States